CLINICAL TRIAL: NCT04420858
Title: Effect of Video Education on Patients' Knowledge and Attitudes of Privacy in Prenatal Genetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1500909-1
Record Dates: First submitted 2020-05-18; First posted 2020-06-09 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Aneuploidy; Genetic Disease; Pregnancy Related
Keywords: Genetic privacy; Aneuploidy screening; Pregnancy; Data use; Data sharing; Protected health information
MeSH Terms: conditions — Aneuploidy; Genetic Diseases, Inborn | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): The control arm will receive standard education about cell-free DNA screening that would typically be presented during a prenatal visit.
  Interventions: Behavioral: Standard (control) education.
- Experimental (Experimental): The experimental arm will receive additional education about federal legislation that protects the privacy of genetic information (Genetic Information Nondiscrimination Act, GINA).
  Interventions: Behavioral: Enhanced (experimental) education

INTERVENTIONS:
Behavioral: Enhanced (experimental) education — See arm description.
  Arms: Experimental
Behavioral: Standard (control) education. — See arm description.
  Arms: Control

SUMMARY:
The investigators propose a randomized controlled trial to assess baseline maternal knowledge of and attitudes toward commercial prenatal genetic testing laboratories' genetic privacy practices, and to determine whether a brief educational intervention alters these attitudes.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial to assess baseline maternal knowledge of and attitudes toward commercial prenatal genetic testing laboratories' genetic privacy practices, and to determine whether a brief educational intervention alters these attitudes. Pregnant women undergoing specialized fetal anatomic ultrasound surveys at Women and Infants' maternal fetal medicine prenatal diagnostic imaging centers will be recruited to participate. Volunteers will be randomized to receive either standard education about prenatal genetic testing or standard education plus additional education about federal genetic privacy protections. Next, the participants view the educational materials to which they were randomized. Finally, all volunteers will take the same survey, which will assess baseline demographic variables as well as their knowledge of and attitudes toward broad sharing of data obtained from prenatal genetic testing. Once finished with the survey, volunteers will have completed their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients undergoing a scheduled L2 ultrasound at the Women and Infants Prenatal Diagnosis Center (PDC)
* Singleton pregnancies
* English speaking
* Results available from cell-free DNA screening for this pregnancy

Exclusion Criteria:

* Prior L2 ultrasound at the PDC during the current pregnancy (to avoid test-retest or multiple approach)
* Prior participation in this study
* Gestational age <17'0 weeks or >23'6 weeks
* Suboptimally dated pregnancies (i.e. dated by ultrasound after 22 weeks gestation)
* Unscheduled / add-on L2 ultrasounds

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Knowledge about broad sharing of genetic data for non-clinical research purposes | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: What is patient knowledge about the potential sharing of their genetic data for non-clinical research purposes? Outcome will be measured on the Likert scale.
Acceptability of broad sharing of genetic data for non-clinical research purposes | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: What is patient acceptance of laboratory-initiated sharing of their de-identified genetic data for non-clinical purposes? Outcome will be measured on the Likert scale.

SECONDARY OUTCOMES:
Acceptability of retention of genetic data for non-clinical purposes | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: What is patient acceptance of retaining their de-identified genetic data to potentially use it for non-clinical purposes? Outcome will be measured on the Likert scale.
Acceptability of use of genetic data for non-clinical purposes | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: What is patient acceptance of using their de-identified genetic data for non-clinical purposes such as research and development? Outcome will be measured on the Likert scale.
Knowledge and understanding of aneuploidy screening and results | This outcome will be assessed immediately after exposure to education (day 0)
  Are patients aware that they underwent aneuploidy screening with cell-free fetal DNA (cfDNA)? Are they aware of their results? Outcome will be measured on the Likert scale.
Knowledge and understanding of carrier testing and results | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: Are patients aware that they underwent carrier testing? Are they aware of their results? Outcome will be measured on the Likert scale.
Acceptability of retention, use, and broad sharing of fetal genetic data for non-clinical research purposes | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: Assess maternal acceptance of each of these outcomes. Outcome will be measured on the Likert scale.
Maternal rationale for pursuing cfDNA | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: What prompted patient to pursue cfDNA testing? Outcome will be measured on the Likert scale.
Maternal knowledge of different commercial cfDNA providers | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: Are patents who have undergone cfDNA testing aware that multiple companies offer this service? Outcome will be measured on the Likert scale.
Maternal knowledge pertaining to Down Syndrome and the genetics of trisomies. | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: To what extent do mothers who have undergone cfDNA screening and are participating in this study understand these topics? Outcome will be measured on the Likert scale.
Maternal perceptions of the de-identifiability of genetic data | This outcome will be assessed immediately after exposure to education (day 0)
  Using a newly designed survey instrument (the Prenatal Testing Opinions Survey), the investigators aim to answer the following question: To what extent do mothers who have undergone cfDNA screening believe that deidentified genetic information is not re-identifiable? Outcome will be measured on the Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Parobek, Principal Investigator — Department of OB/GYN, Women and Infants Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable data will be freely shared with other researchers upon request for facilitate reproducibility or future systemic review, pending approval from local institutional review board.
Time Frame: De-identified study data will be available after publication and for a time period of 6 years after enrollment of the final volunteer.
Access Criteria: De-identified study data will be shared with researchers upon request.

REFERENCES:
- [Derived] Parobek CM, Thorsen MM, Has P, Lorenzi P, Clark MA, Russo ML, Lewkowitz AK. Video education about genetic privacy and patient perspectives about sharing prenatal genetic data: a randomized trial. Am J Obstet Gynecol. 2022 Jul;227(1):87.e1-87.e13. doi: 10.1016/j.ajog.2022.03.047. Epub 2022 Mar 26. PMID 35351406
- [Derived] Parobek CM, Has P, Lorenzi P, Russo ML, Clark MA, Lewkowitz AK. What test did I have? Patient uncertainty about prenatal genetic screening. Am J Obstet Gynecol. 2021 Sep;225(3):341-342. doi: 10.1016/j.ajog.2021.05.030. Epub 2021 May 27. No abstract available. PMID 34051169